CLINICAL TRIAL: NCT04775914
Title: The STEMI Optimization Trial - Ischemic Postconditioning (DANAMI4-iPOST) and Intravascular Ultrasound Guided PCI in STEMI (DANAMI4-iSTEMI)
Brief Title: STEMI Treatment Optimization by Ischemic Postconditioning and IVUS Guidance
Acronym: DANAMI4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Engstrom (Other)
Responsible Party: Sponsor-Investigator, Thomas Engstrom, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H-18051256b
Record Dates: First submitted 2021-02-17; First posted 2021-03-01 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Primary PCI; Coronary angiography; Intravascular ultra sound (IVUS)
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Stents; High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: 2x2 factorial
  As a second randomization to the iPOST2 trial (ID: H-180512561,NCT03787745) patients are randomized 1:1 to either a) receiving ultrasound guidance before and after stent placement or b) no ultrasound, independently of randomization in the iPOST2 trial. The iPOST2 trial was initiated February 2019.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PCI standard (Active Comparator)
  Interventions: Procedure: PCI + Ischemic conditioning
- PCI standard + ischemic conditioning (Experimental)
  Interventions: Procedure: PCI + Ischemic conditioning
- Stent with ultrasound (Experimental)
  Interventions: Procedure: Stent with ultrasound
- Stent without ultrasound (Active Comparator)
  Interventions: Procedure: Stent with ultrasound

INTERVENTIONS:
Procedure: PCI + Ischemic conditioning — IPOST is repeated for 4 cycles (60 sec obstruction followed by 60 sec perfusion each) and followed by stent implantation with a 1.1/1.0 ratio of stent diameter/reference vessel diameter and a stent length sufficient to cover the entire lesion from healthy to healthy area of the vessel. During the first cycle of re-occlusion of full vessel occlusion is secured by a small injection of contrast.
  Arms: PCI standard; PCI standard + ischemic conditioning
Procedure: Stent with ultrasound — IVUS catheters are to be advanced at least 20 mm distal to the culprit lesion. After administration of intracoronary nitroglycerine, an IVUS-pullback is to be performed at 0.5mm/second using a commercially available imaging system. Stent size and landing zones are decided based on the IVUS.
  Arms: Stent with ultrasound; Stent without ultrasound

SUMMARY:
The purpose of is study is to investigate whether ischemic postconditioning (iPOST) and intravascular ultrasound-guided (IVUS) percutaneous coronary intervention (PCI) improve the clinical outcome of patients with ST-segment elevation myocardial infarction treated with primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute onset of chest pain with <12 hours duration
* STEMI as characterized by 2 mm ST elevation in 2 or more V1 through V4 leads or presumed new left bundle branch block with minimum of 1 mm concordant ST elevation or 1 mV ST-segment elevation in the limb lead (II, III and aVF, I, aVL) and V4-V6 or ST depression in 2 or more V1 through V4 leads indicating posterior AMI.

Exclusion Criteria (iPOST2):

Pre-PCI TIMI flow 0 or 1 Potential pregnancy Inability to provide informed consent Unwillingness to consent Unavoidable to use thrombectomy Spontaneous coronary artery dissection Time from symptoms onset to PPCI > 12 hours Culprit in bypass graft Other reason for not including the patient

Exclusion Criteria (iSTEMI):

Potential pregnancy Inability to understand information in order to provide informed consent Unwillingness to consent Spontaneous coronary artery dissection Time from symptoms inset to PPCI > 12 hours Culprit in bypass graft Other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
iPOST | Until expected number of events are adjudicated up til 3 years
  Number of participants that experience all-cause mortality or hospitalization for heart failure
iSTEMI (IVUS) | Until expected number of events are adjudicated up til 3 years
  Number of participants that experience all-cause mortality, unplanned ischemia-driven revascularization and new myocardial infarction

SECONDARY OUTCOMES:
iSTEMI (IVUS) | Until expected number of events are adjudicated 3 years
  Target vessel failure (cardiac mortality, unplanned ischemia driven target vessel revascularization or target vessel myocardial infarction
iSTEMI (IVUS) | Until expected number of events are adjudicated 3 years
  Individual components of the primary endpoint
iSTEMI (IVUS) | Until expected number of events are adjudicated 3 years
  Cardiac mortality
iSTEMI (IVUS) | Until expected number of events are adjudicated 3 years
  Unplanned ischemia driven target vessel revascularization
iSTEMI (IVUS) | Until expected number of events are adjudicated 3 years
  Unplanned ischemia driven target vessel myocardial infarction
iSTEMI (IVUS) | Until expected number of events are adjudicated 3 years
  Unplanned ischemia driven target lesion revascularization
iSTEMI (IVUS) | Until expected number of events are adjudicated 3 years
  Definite/probable stent-thrombosis
iPOST | Until expected number of events are adjudicated 3 years
  Individual components of the primary endpoint
iPOST | Until expected number of events are adjudicated 3 years
  Cardiac mortality
iPOST | Until expected number of events are adjudicated 3 years
  Ischemia driven target vessel revascularization
iPOST | Until expected number of events are adjudicated 3 years
  New myocardial infarction
iPOST | 1 year
  Quality of life

OTHER OUTCOMES:
iSTEMI (IVUS) | Until expected number of events are adjudicated 3 years
  Hospitalization for heart failure
iSTEMI (IVUS) | Until expected number of events are adjudicated 3 years
  Stroke
iSTEMI (IVUS) | Until expected number of events are adjudicated 3 years
  Bleeding
iSTEMI (IVUS) | 1 year
  Quality of life
iPOST | Until expected number of events are adjudicated 3 years
  Any ischemia driven revascularization
iPOST | Until expected number of events are adjudicated 3 years
  Bleeding
iPOST | Until expected number of events are adjudicated 3 years
  Stroke
iPOST | Until expected number of events are adjudicated 3 years
  Ventricular arrythmia
iPOST | Until expected number of events are adjudicated 3 years
  ICD

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Engstrøm, MD PhD DMSci, Study Chair — Rigshospitalet, Denmark; Jacob Lønborg, MD PhD DMSci, Study Chair — Rigshospitalet, Denmark; Francis Joshi, Md, PhD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Heart Center, Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No